CLINICAL TRIAL: NCT05535478
Title: Deprescribing of Diabetes Treatment Regimens in Long Term Care (LTC) Residents With Alzheimer's Disease or Related Dementias (ADRD)
Brief Title: Deprescribing of Diabetes Regimens in Long Term Care Residents With Alzheimer's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Brown University (Other); Theoria Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00053280
Record Dates: First submitted 2022-08-26; First posted 2022-09-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Diabetes; Dementia; Hypoglycemia; Drug
Keywords: older adults; long term care facility; high risk medications; hypoglycemia; deprescribing; diabetes; dementia
MeSH Terms: conditions — Diabetes Mellitus; Dementia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- STRIDE Intervention (Other): Educational intervention for clinicians
  Interventions: Behavioral: STRIDE

INTERVENTIONS:
Behavioral: STRIDE — a. Targeted providers for STRIDE program: i. Clinical staff at the LTCF who participate in deprescribing at the facilities (physicians (MDs), physician's assistants (PAs), nurse practitioners (NPs), clinical pharmacists): clinical staff members caring for LTCF residents with ADRD and diabetes at 6 LTCFs in the Ohio and Michigan areas will be invited via email from the LTCF leadership to participate in the STRIDE education program. The STRIDE program consist of practical algorithms and educational material, which they are free to view at any time, and participation in 2 webinars and monthly telementoring calls

SUMMARY:
Objectives To 1) examine the ability of the STRIDE (Simplification of Treatment Regimens and Individualized Diabetes Education) educational program to increase deprescribing of high hypoglycemia risk glucose-lowering medications (HRMs) among long term care facility (LTCF) residents with ADRD, 2) assess key implementation constructs (secondary outcomes) of the STRIDE program, including acceptability, appropriateness, and feasibility, and 3) validate the primary HRM use outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical staff at the LTCF (MDs, PAs, NPs, clinical pharmacists) - (Targeted providers for STRIDE program)
* Clinical staff that participated in the STRIDE program (Providers doing stakeholder exit interviews)

Exclusion Criteria:

* Consistent with the pragmatic nature of the trial, there are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Change in proportion of long term care facility (LTCF) residents with Alzheimer's disease adn related dementias (ADRD) and diabetes with high risk medications (HRM) use | Baseline vs 6 months
  HRM use will include any sulfonylurea use (i.e., glyburide, glipizide, glimepiride, or chlorpropamide) and any insulin use.

SECONDARY OUTCOMES:
Acceptability of the STRIDE Educational Program | 6 months
  The extent to which the program is agreeable to LTCF staff- using the Acceptability of Intervention Measure (AIM)
Appropriateness of the STRIDE Educational Program | 6 months
  The extent to which the program is suitable for a particular purpose, i.e., to improve the frequency at which LTCF staff attempt diabetes medication regimen deprescribing- using the Intervention Appropriateness Measure (IAM)
Feasibility of the STRIDE Educational Program | 6 months
  The extent to which the program is practical at the LTCF level- using the Feasibility of Intervention Measure (FIM)

CONTACTS AND LOCATIONS:
Overall Officials: Medha Munshi, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No